CLINICAL TRIAL: NCT01760265
Title: Dysbetalipoproteinemia and Atheroma Risk : Assessment of Cardiovascular Risk in Dysbetalipoproteinemic Patients
Brief Title: DARK STUDY "DysbetalipoproteinemiA and atheRoma Risk"
Acronym: DARK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Dysbetalipoproteinemia
Keywords: dysbetalipoproteinemia; artery calcium score; carotid intima media; ankle brachial index; dysbetalipoproteinemic patients
MeSH Terms: conditions — Hyperlipoproteinemia Type III

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Lipid, apo E genotype when is necessary to complete the phenotype
Oversight: Data Monitoring Committee: No

SUMMARY:
Dysbetalipoproteinemia (type III, Fredrickson's classification) is a rare metabolic disorder. It results from a defect in the clearance of VLDL and chylomicron remnants due to homozygous APOE2 variants or heterozygous APOE mutations, and there is an elevated plasma cholesterol and triglycerides.

As a consequence of the derangements in lipoprotein metabolism, dysbetalipoproteinemia predispose to the premature development of atherosclerosis.

However among this population there is heterogeneity in development of cardiovascular complications and the determinants remain unclear actually.

The aim of the investigators study is to evaluate the intensity of clinical atherosclerosis, and identify its determinants.

ELIGIBILITY:
Inclusion Criteria:

- apo E gene sequencing in CBE (Centre de Biologie Est / Hospices Civils de Lyon / France) laboratory in Lyon until December 2012

Exclusion Criteria:

* age < 40 years
* refused participation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dysbetalipoproteinemia patients with APOE2/E2 or heterozygous mutation (negative dominance) and hypercholesterolemia, ratio CT VLDL/Tg VLDL >0.40
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Computed tomographic measurements for coronary-artery calcium | Day one : the coronary calcium score is assessed on the date of measurement
  Comparison with eventual previous examinations.

SECONDARY OUTCOMES:
Measurement of carotid intima-media by ultrasonography | Day one : on the date of measurement
  Comparison with eventual previous examinations.
Measurement of ankle brachial index | Day one : on the date of measurement
  Comparison with eventual previous examinations

CONTACTS AND LOCATIONS:
Overall Officials: Philippe MOULIN, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon - Groupement Hospitalier Est, Bron, France